CLINICAL TRIAL: NCT01421043
Title: An Open Label, Randomized, Single Dose, Crossover Pivotal Bioequivalence Study of Triazolam Liquid Oral Drops at a Dose of 0.25 Mg Versus Triazolam 0.25 Mg Tablet in Healthy Subjects
Brief Title: A Study to Determine Whether an Oral Drops Formulation of Triazolam is Bioequivalent to a Tablet Formulation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6781003
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: bioequivalence study; triazolam; liquid oral drops; tablet
MeSH Terms: interventions — Triazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- triazolam liquid oral drops (Experimental)
  Interventions: Drug: triazolam liquid oral drops
- triazolam tablets (Active Comparator)
  Interventions: Drug: triazolam tablets

INTERVENTIONS:
Drug: triazolam liquid oral drops — 0.25 mg single dose oral drops
  Arms: triazolam liquid oral drops
Drug: triazolam tablets — 0.25 mg single oral dose
  Arms: triazolam tablets

SUMMARY:
This study will determine whether an oral drops formulation of triazolam at a dose of 0.25 mg is bioequivalent to a tablet formulation at a dose of 0.25 mg in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) to last time point (t) | 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16 and 24 hours postdose
Maximum concentration of drug (Cmax) | 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16 and 24 hours postdose

SECONDARY OUTCOMES:
Area Under the Curve (AUC) to time infinity (inf) (if data permit) | 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16 and 24 hours postdose
Area Under the Curve (AUC) percent extrapolated (%exp) | 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16 and 24 hours postdose
Half-life (if data permit) | 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16 and 24 hours postdose
Time at maximum concentration (Tmax) | 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16 and 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6781003&StudyName=A%20Study%20to%20Determine%20Whether%20an%20Oral%20Drops%20Formulation%20of%20Triazolam%20is%20Bioequivalent%20to%20a%20Tablet%20Formulation%20in%20Healthy%20Subjects